CLINICAL TRIAL: NCT02895841
Title: Patient-Empowered Mobile Technology in Hospitalized Patients: Technology Resources to Understand Pain Assessment in Patients With Pain (TRU-PAIN)
Brief Title: Patient-Empowered Mobile Technology in Hospitalized Patients (TRU-PAIN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00068979
Record Dates: First submitted 2016-09-01; First posted 2016-09-12 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Pain
Keywords: oncology; bone marrow transplant; sickle cell disease
MeSH Terms: conditions — Pain; Neoplasms; Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Patients will continue with their normal Standard of Care for their condition
- SMART app wearable device (Experimental): Patients will be given a wearable such as a Microsoft Band accelerometer to track movement, heart rate, galvanic skin response and sleep, which will be collected in combination with the data from the SMART visual dashboard. Data will be sent to the SMART dashboard as well as stored on the iPad/iPod touch via software from the manufacturer. Participants having a "wearable device" will receive the education intervention (such as haptic prompted texts that state 'try and walk today', 'have you had enough water today', 'make sure to take deep breaths').
  Interventions: Other: SMART app wearable

INTERVENTIONS:
Other: SMART app wearable — Patients will be given a wearable such as a Microsoft Band accelerometer to track movement, heart rate, galvanic skin response and sleep, which will be collected in combination with the data from the SMART visual dashboard. Data will be sent to the SMART dashboard as well as stored on the iPad/iPod touch via software from the manufacturer. Participants having a "wearable device" will receive the education intervention (such as haptic prompted texts that state 'try and walk today', 'have you had enough water today', 'make sure to take deep breaths').
  Arms: SMART app wearable device

SUMMARY:
The purpose of this study is to learn more about the ways in which mobile technology can be integrated into inpatient care to help better track pain levels using mobile technology of patients with sickle cell disease, oncology patients, and bone marrow transplant patients. The study will assess whether or not daily mobile monitoring with wearable accelerometers (devices that detect movement as well as heart-rate) to monitor and manage medical treatments can have a lasting positive impact on outcomes in patients with chronic diseases. The investigator hopes to learn more about the ways in which mobile technology can be integrated into inpatient care. Specifically, the investigator is looking to help patients better track their pain, use wearable technology to track physiological measures (for example, heart rate, sleep quantity and quality), and integrate these data points into the medical care of patients by providing the information to providers. This study will first gather information regarding the feasibility and acceptability of the use of technology on the inpatient unit. This will help the study team to refine the technology of the mobile app and logistics of integration. Following this, the investigator will complete a second phase of the study, during which select patients will pilot the intervention. This will be followed by the third and final phase, during which patients will be randomly assigned to the active intervention or standard of care. This phase approach will enable the study team to refine the intervention, relying on the feedback from patients and providers, and subsequently test its utility compared to standard of care through random assignment.

DETAILED DESCRIPTION:
The investigator hopes to learn more about the ways in which mobile technology can be integrated into inpatient care. Specifically, the investigator is looking to help patients better track their pain, use wearable technology to track physiological measures (for example, heart rate, sleep quantity and quality), and integrate these data points into the medical care of patients by providing the information to providers. This study will first gather information regarding the feasibility and acceptability of the use of technology on the inpatient unit. This will help the study team to refine the technology of the mobile app and logistics of integration. Following this, the investigator will complete a second phase of the study, during which select patients will pilot the intervention. This will be followed by the third and final phase, during which patients will be randomly assigned to the active intervention or standard of care. This phase approach will enable the study team to refine the intervention, relying on the feedback from patients and providers, and subsequently test its utility compared to standard of care through random assignment.

ELIGIBILITY:
Inclusion Criteria:

* Any patient 8-80 years old with a past medical history for a chronic disease (such as sickle cell disease), cancer (solid tumor, lymphoma, brain tumor), or currently undergoing bone marrow transplant
* Currently admitted to the hospital
* Have a current diagnosis which includes pain for which they are being treated

Exclusion Criteria:

* Must be enrolled within 48 hours of admission
* Due to the possibility of a choking hazard, only patients who are at least 8 years of age will be enrolled in the study
* Patients in the Intensive Care Units will not be eligible
* Must be able to understand and operate the mobile device independently; therefore the investigators will exclude those the provider team considers unable to do so

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2016-08; Primary Completion 2024-04-22 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
time to discontinuation of the IV PCA with opioid medication | 7 days

SECONDARY OUTCOMES:
time of movement during hospitalization | 7 days
magnitude of change in pain scores | 7 days
patient/family satisfaction scores as measured by feasibility survey | 7 days
  A 24-item survey was developed for parents and children assessing technical feasibility, adherence

CONTACTS AND LOCATIONS:
Overall Officials: Nirmish Shah, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaughn J, Gollarahalli S, Shaw RJ, Docherty S, Yang Q, Malhotra C, Summers-Goeckerman E, Shah N. Mobile Health Technology for Pediatric Symptom Monitoring: A Feasibility Study. Nurs Res. 2020 Mar/Apr;69(2):142-148. doi: 10.1097/NNR.0000000000000403. PMID 31972852